CLINICAL TRIAL: NCT00617305
Title: An Open-label, Multicenter Study of Ambrisentan and a Phosphodiesterase Type-5 Inhibitor Combination Therapy in Subjects With Pulmonary Arterial Hypertension Who Have Demonstrated a Sub-Optimal Response to a Phosphodiesterase Type-5 Inhibitor
Brief Title: Study of Add-on Ambrisentan Therapy to Background Phosphodiesterase Type-5 Inhibitor (PDE5i) Therapy in Pulmonary Arterial Hypertension (ATHENA-1)
Acronym: ATHENA-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-US-300-0117
Record Dates: First submitted 2008-02-06; First posted 2008-02-18 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-06

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: ambrisentan; PAH; combination therapy; phosphodiesterase type-5 inhibitor (PDE-5i); cardiovascular; endothelin receptor antagonist; ERA
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ambrisentan; Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan (Experimental): Patients were assigned ambrisentan at open-label enrollment or randomization, and received at least one dose of ambrisentan plus an approved phosphodiesterase type-5 (PDE-5) inhibitor (PDE-5i; sildenafil or tadalafil).
  Interventions: Drug: Ambrisentan; Drug: Sildenafil; Drug: Tadalafil
- Placebo (Active Comparator): Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i (sildenafil or tadalafil).
  Interventions: Drug: Placebo; Drug: Sildenafil; Drug: Tadalafil

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan was administered orally once daily; dose level was 5 mg for the first 4 weeks, followed by 10 mg for the remainder of the study; ambrisentan was supplied as 5-mg and 10-mg tablets.
  Other Names: Letairis
  Arms: Ambrisentan
Drug: Placebo — Placebo to match ambrisentan was administered orally once daily.
  Arms: Placebo
Drug: Sildenafil — Sildenafil was administered at the dose previously established for each subject (20-100 mg) orally three times daily. Sildenafil was supplied as 20-mg tablets, or formulated as sildenafil citrate in 25-, 50-, or 100-mg tablets.
  Other Names: Revatio; Viagra
Drug: Tadalafil — Tadalafil was administered at the dose previously established for each subject (not to exceed 40 mg per day) orally once daily. Tadalafil was supplied as 20-mg tablets.
  Other Names: Cialis; Adcirca

SUMMARY:
To evaluate the change from baseline in pulmonary vascular resistance (PVR), and other hemodynamic parameters, following the addition of ambrisentan to background phosphodiesterase type-5 inhibitor (PDE-5i) therapy in subjects with pulmonary arterial hypertension (PAH) who have demonstrated a sub-optimal response to PDE-5i monotherapy.

The study was originally designed as a 2-arm, double-blind, randomized study in which patients received ambrisentan or placebo for 24 weeks, and then received ambrisentan blinded to dose for 24 weeks. With Protocol Amendment 2 (12 June, 2009), the study was switched to single-arm, open-label treatment, and all patients remaining in the placebo arm were switched to open-label ambrisentan treatment. Patients who enrolled after Amendment 2 all received open-label ambrisentan.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the change from baseline in pulmonary vascular resistance (PVR), and other hemodynamic parameters, following the addition of ambrisentan to background phosphodiesterase type-5 inhibitor (PDE-5i) therapy in subjects with pulmonary arterial hypertension (PAH) who have demonstrated a sub-optimal response to PDE-5i monotherapy.

The secondary objectives of this study are to evaluate the change from baseline in other clinical measures of PAH following the addition of ambrisentan to background PDE-5i therapy in subjects with PAH who have demonstrated a sub-optimal response to PDE-5i monotherapy.

The safety and tolerability of ambrisentan/PDE-5i combination therapy will be evaluated throughout the study. In addition, long-term efficacy will be examined.

ELIGIBILITY:
Selected Inclusion Criteria

* Must be between 16 and 75 years of age;
* Must weigh at least 40 kg;
* Have a current diagnosis of idiopathic PAH, familial PAH, or PAH that is primarily due to connective tissue disease, congenital heart defects, drug or toxin use, or human immunodeficiency virus (HIV);
* Have WHO functional class III symptoms;
* Be receiving sildenafil or tadalafil monotherapy for the treatment of PAH for at least the past 12 weeks and at a stable dose for at least 8 consecutive weeks;
* Meet all of the following hemodynamic criteria by means of a right heart catheterization: mPAP of at least 25 mmHg; PVR of at least 400 dyne*sec/cm5; pulmonary capillary wedge pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) of not more than 15 mmHg;
* Meet all of the following pulmonary function test criteria no more than 12 weeks before the screening visit: total lung capacity at least 60% of predicted normal and forced expiratory volume in 1 second of at least 65% of predicted normal;
* Able to walk at least 150 meters during the screening 6-minute walk test (6MWT);
* If receiving calcium channel blockers or 5-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors (i.e., statins) must be on stable therapy for at least 4 weeks;
* If diagnosed with HIV, must have stable disease status.

Selected Exclusion Criteria:

* Have a current pulmonary hypertension diagnosis other than idiopathic PAH, familial PAH, or PAH that is primarily due to connective tissue disease, congenital heart defects, drug or toxin use, or HIV;
* Have left ventricular ejection fraction (LVEF) ≤40% or clinically significant ischemic, valvular, or constrictive heart disease;
* Have received chronic prostanoid or endothelin receptor antagonist (ERA) therapy (eg, bosentan, sitaxsentan) within the past 12 weeks;
* Have discontinued ERA treatment for any adverse reaction other than those associated with liver function test abnormalities;
* Have received IV inotropes within 2 weeks;
* Have a serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value that is greater than 2.0x the upper limit of normal.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - University of South Alabama, Mobile, Alabama
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - West Los Angeles Healthcare Center, Los Angeles, California
  - Harbor - UCLA, Torrance, California
  - Cleveland Clinic, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Heart Center, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - University of Iowa, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - BACH Cardiology, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Cornell Medical Center, New York, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Scott & White Memorial Hospital, Temple, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

REFERENCES:
- See also: Click here for more information about ambrisentan — http://www.letairis.com/patients/default.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled in 16 study sites in the US. The first patient was screened on 09 April 2008, and the last patient was enrolled on 28 July 2010. The last patient observation was on 25 July 2011. Originally a double-blind, placebo-controlled study, it was changed to open label on 12 June 2009 due to slow enrollment.
Pre-assignment Details: 65 patients were screened; 8 were randomized (3 to ambrisentan and 5 to placebo) prior to study conversion to open label. The remaining patients were assigned to ambrisentan treatment.
Groups:
- Ambrisentan Only: Patients were assigned ambrisentan at open-label enrollment or randomization, and received at least one dose of ambrisentan plus an approved phosphodiesterase type-5 (PDE-5) inhibitor (PDE-5i)
- Placebo/Ambrisentan: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i; patients also received at least one dose of open-label ambrisentan plus an approved PDE-5i
- Placebo Only: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i
Period: Overall Study
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only
Started | 33 | 4 | 1
Completed 24-week Primary Analysis | 31 | 4 | 0
Completed | 25 | 4 | 0
Not Completed | 8 | 0 | 1
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Total
Number analyzed (Participants) | 33 | 4 | 1 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 4 | 1 | 34
  >=65 years | 4 | 0 | 0 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 48.2 (13.72) | 43.5 (14.89) | 49.0 (0) | 47.8 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 2 | 0 | 28
  Male | 7 | 2 | 1 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 0 | 8
  Not Hispanic or Latino | 25 | 4 | 1 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2 | 0 | 0 | 2
  Black or African American | 2 | 0 | 0 | 2
  Hispanic | 1 | 0 | 0 | 1
  More than one race | 1 | 0 | 0 | 1
  White | 27 | 4 | 1 | 32
Region of Enrollment [Number; unit: participants]
  United States | 33 | 4 | 1 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pulmonary Vascular Resistance (PVR), Last Observation Carried Forward (LOCF)
Description: The primary objective of this study is to evaluate the change from baseline in PVR, and other hemodynamic parameters, following the addition of ambrisentan to background PDE-5i therapy in subjects with PAH who have demonstrated a sub-optimal response to PDE-5i monotherapy. A decrease in measurement value (dynes sec/cm^5) indicates improvement for this patient population.
Time Frame: Baseline to Week 24
Population: Patients with measurements at Baseline and Week 24 were evaluated
Measure: Mean (Standard Deviation); unit: dynes sec/cm^5
Groups:
- Ambrisentan Only: Patients were assigned ambrisentan at open-label enrollment or randomization, and received at least one dose of ambrisentan plus an approved phosphodiesterase type-5 (PDE-5) inhibitor (PDE-5i) (33 patients had baseline measurements in this group)
- Placebo/Ambrisentan: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i; patients also received at least one dose of open-label ambrisentan plus an approved PDE-5i (4 patients had baseline measurements in this group)
- Placebo Only: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i and did not receive ambrisentan (1 patient had baseline measurements in this group)
- Any Ambrisentan: Patients were assigned either ambrisentan or placebo at enrollment or randomization and received at least one dose of ambrisentan plus an approved PDE-5i (37 patients had baseline measurements in this group)
- Any Placebo: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i (5 patients had baseline measurements in this group)
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 31 | 4 | 0 | 35 | 4
dynes sec/cm^5
  Baseline | 761.2 (306.57) | 731.6 (278.02) |  | 758.0 (300.12) | 703.6 (248.73)
  Week 24 | 518.8 (196.35) | 439.8 (130.34) |  | 509.8 (190.18) | 439.8 (130.34)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -248.93, 95% CI 2-sided [-337.7 to -160.2], Standard Deviation 241.978
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -291.80, 95% CI 2-sided [-619.4 to 35.78], Standard Deviation 205.864
Statistical Analysis 3: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -253.83, 95% CI 2-sided [-334.8 to -172.8], Standard Deviation 235.787
Statistical Analysis 4: Comparison: Any Placebo; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -291.80, 95% CI 2-sided [-619.4 to 35.78], Standard Deviation 205.864

2. Secondary Outcome: Change From Baseline in Mean Pulmonary Artery Pressure (mPAP) (LOCF)
Description: This secondary hemodynamic outcome is supportive of the primary outcome. A decrease in measurement value (mmHg) indicates improvement for this patient population.
Time Frame: Baseline to Week 24
Population: Patients with measurements at Baseline and Week 24 were evaluated
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 31 | 4 | 0 | 35 | 4
mmHg
  Baseline | 49.9 (9.75) | 54.5 (12.50) |  | 50.4 (9.98) | 52.8 (11.48)
  Week 24 | 44.4 (10.95) | 38.8 (9.60) |  | 43.8 (10.83) | 38.8 (9.60)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -5.38, 95% CI 2-sided [-8.29 to -2.46], Standard Deviation 7.954
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -15.75, 95% CI 2-sided [-29.64 to -1.86], Standard Deviation 8.732
Statistical Analysis 3: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -6.56, 95% CI 2-sided [-9.51 to -3.61], Standard Deviation 8.589
Statistical Analysis 4: Comparison: Any Placebo; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -15.75, 95% CI 2-sided [-29.64 to -1.86], Standard Deviation 8.732

3. Secondary Outcome: Change From Baseline in Mean Right Atrial Pressure (mRAP) (LOCF)
Description: as for outcome 2
Time Frame: Baseline to Week 24
Population: Patients with measurements at Baseline and Week 24 were evaluated
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 31 | 4 | 0 | 35 | 4
mmHg
  Baseline | 8.5 (4.82) | 10.3 (2.63) |  | 8.7 (4.64) | 11.1 (2.97)
  Week 24 | 8.4 (4.88) | 6.3 (1.71) |  | 8.1 (4.66) | 6.3 (1.71)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -0.06, 95% CI 2-sided [-1.69 to 1.56], Standard Deviation 4.442
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -4.00, 95% CI 2-sided [-10.50 to 2.50], Standard Deviation 4.082
Statistical Analysis 3: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -0.51, 95% CI 2-sided [-2.07 to 1.04], Standard Deviation 4.527
Statistical Analysis 4: Comparison: Any Placebo; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = -4.00, 95% CI 2-sided [-10.50 to 2.50], Standard Deviation 4.082

4. Secondary Outcome: Change From Baseline in Cardiac Output (LOCF)
Description: This secondary hemodynamic outcome is supportive of the primary outcome. An increase in measurement value (L/min) indicates improvement for this patient population.
Time Frame: Baseline to Week 24
Population: Patients with measurements at Baseline and Week 24 were evaluated
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 28 | 4 | 0 | 32 | 4
L/min
  Baseline | 4.4 (1.22) | 4.8 (0.81) |  | 4.4 (1.17) | 4.8 (0.71)
  Week 24 | 5.2 (1.27) | 5.2 (1.22) |  | 5.2 (1.24) | 5.2 (1.22)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = 0.84, 95% CI 2-sided [0.43 to 1.25], Standard Deviation 1.053
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.77 to 1.42], Standard Deviation 0.685
Statistical Analysis 3: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = 0.78, 95% CI 2-sided [0.41 to 1.15], Standard Deviation 1.021
Statistical Analysis 4: Comparison: Any Placebo; Mean change from Baseline to Week 24; Test type: Superiority or Other; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.77 to 1.42], Standard Deviation 0.685

5. Secondary Outcome: Change From Baseline in Six Minute Walk Distance (6MWD) Measured at Weeks 4, 12, 24, 36 and 48 (LOCF)
Description: The primary analysis of this secondary outcome measure is mean change from Baseline to Week 24. The changes from Baseline to Weeks 4, 12, 36, and 48 were also evaluated. An increase in measurement value (meters walked) indicates improvement for this patient population.
Time Frame: Baseline to Week 48
Population: All enrolled Population
Measure: Mean (Standard Deviation); unit: meters walked
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 33 | 4 | 1 | 37 | 5
meters walked
  Baseline | 361.9 (98.74) | 433.3 (80.77) | 335.0 (0.0) | 369.6 (98.56) | 413.6 (82.61)
  Week 4 | 376.5 (106.08) | 441.0 (83.88) | 442.0 (0.0) | 383.7 (104.85) | 441.2 (72.65)
  Week 12 | 377.9 (109.61) | 435.8 (134.61) | 422.0 (0.0) | 384.3 (111.96) | 433.0 (116.74)
  Week 24 | 382.4 (104.96) | 423.8 (110.05) | 422.0 (0.0) | 387.0 (104.73) | 423.4 (95.31)
  Week 36 | 366.5 (127.62) | 399.3 (152.93) | 402.0 (0.0) | 370.2 (128.61) | 399.8 (132.45)
  Week 48 | 378.9 (124.18) | 383.5 (192.47) | 402.0 (0.0) | 379.4 (129.75) | 387.2 (166.89)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 12.2, 95% CI 2-sided [-3.9 to 28.4], Standard Deviation 44.84
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 7.8, 95% CI 2-sided [-26.0 to 41.5], Standard Deviation 21.19
Statistical Analysis 3: Comparison: Placebo Only; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 107.0, Standard Deviation 0.0
Statistical Analysis 4: Comparison: Any Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 11.7, 95% CI 2-sided [-2.7 to 26.2], Standard Deviation 42.68
Statistical Analysis 5: Comparison: Any Placebo; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 27.6, 95% CI 2-sided [-32.0 to 87.2], Standard Deviation 48.03
Statistical Analysis 6: Comparison: Ambrisentan Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 13.6, 95% CI 2-sided [-1.4 to 28.5], Standard Deviation 41.46
Statistical Analysis 7: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 2.5, 95% CI 2-sided [-91.5 to 96.5], Standard Deviation 59.09
Statistical Analysis 8: Comparison: Placebo Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 87.0, Standard Deviation 0.0
Statistical Analysis 9: Comparison: Any Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 12.4, 95% CI 2-sided [-2.1 to 26.9], Standard Deviation 42.83
Statistical Analysis 10: Comparison: Any Placebo; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 19.4, 95% CI 2-sided [-59.6 to 98.4], Standard Deviation 63.61
Statistical Analysis 11: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 18.1, 95% CI 2-sided [0.5 to 35.6], Standard Deviation 48.67
Statistical Analysis 12: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -9.5, 95% CI 2-sided [-56.5 to 37.5], Standard Deviation 29.56
Statistical Analysis 13: Comparison: Placebo Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 87.0, Standard Deviation 0.0
Statistical Analysis 14: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 15.0, 95% CI 2-sided [-1.0 to 31.1], Standard Deviation 47.44
Statistical Analysis 15: Comparison: Any Placebo; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 9.8, 95% CI 2-sided [-52.5 to 72.1], Standard Deviation 50.18
Statistical Analysis 16: Comparison: Ambrisentan Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 2.2, 95% CI 2-sided [-25.6 to 30.1], Standard Deviation 77.24
Statistical Analysis 17: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -34.0, 95% CI 2-sided [-182.2 to 114.2], Standard Deviation 93.16
Statistical Analysis 18: Comparison: Placebo Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 67.0, Standard Deviation 0.0
Statistical Analysis 19: Comparison: Any Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.8, 95% CI 2-sided [-28.4 to 24.8], Standard Deviation 78.50
Statistical Analysis 20: Comparison: Any Placebo; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -13.8, 95% CI 2-sided [-128.6 to 101.0], Standard Deviation 92.46
Statistical Analysis 21: Comparison: Ambrisentan Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 14.6, 95% CI 2-sided [-15.0 to 44.2], Standard Deviation 82.07
Statistical Analysis 22: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -49.8, 95% CI 2-sided [-251.4 to 151.9], Standard Deviation 126.75
Statistical Analysis 23: Comparison: Placebo Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 67.0, Standard Deviation 0.0
Statistical Analysis 24: Comparison: Any Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 7.4, 95% CI 2-sided [-22.4 to 37.3], Standard Deviation 88.11
Statistical Analysis 25: Comparison: Any Placebo; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -26.4, 95% CI 2-sided [-177.3 to 124.5], Standard Deviation 121.55

6. Secondary Outcome: Change in Dyspnea Index Measured at Weeks 4, 12, 24, 36 and 48 (LOCF)
Description: The primary analysis of this secondary outcome measure is mean change from Baseline to Week 24. The changes from Baseline to Weeks 4, 12, 36, and 48 were also evaluated. The dyspnea index measures the degree of breathlessness after completion of the 6MWT using a scale of 0 to 10, with 0 indicating no breathlessness and 10 indicating maximum breathlessness.
Time Frame: Baseline to Week 48
Population: All enrolled Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 33 | 4 | 1 | 37 | 5
units on a scale
  Baseline | 3.7 (2.07) | 2.5 (1.29) | 3.0 (0.0) | 3.6 (2.03) | 2.6 (1.14)
  Week 4 | 3.2 (1.68) | 3.3 (2.22) | 2.0 (0.0) | 3.2 (1.71) | 3.0 (2.00)
  Week 12 | 3.2 (1.94) | 4.0 (2.83) | 3.0 (0.0) | 3.3 (2.02) | 3.8 (2.49)
  Week 24 | 2.9 (1.96) | 1.9 (1.31) | 3.0 (0.0) | 2.8 (1.91) | 2.1 (1.24)
  Week 36 | 3.2 (2.29) | 3.5 (2.65) | 3.0 (0.0) | 3.2 (2.29) | 3.4 (2.30)
  Week 48 | 3.1 (2.32) | 3.5 (4.04) | 3.0 (0.0) | 3.1 (2.49) | 3.4 (3.51)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.1 to 0.0], Standard Deviation 1.50
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.8, 95% CI 2-sided [-1.6 to 3.1], Standard Deviation 1.50
Statistical Analysis 3: Comparison: Placebo Only; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.0, Standard Deviation 0.0
Statistical Analysis 4: Comparison: Any Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.9 to 0.1], Standard Deviation 1.54
Statistical Analysis 5: Comparison: Any Placebo; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.4, 95% CI 2-sided [-1.5 to 2.3], Standard Deviation 1.52
Statistical Analysis 6: Comparison: Ambrisentan Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.1 to 0.0], Standard Deviation 1.45
Statistical Analysis 7: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 1.5, 95% CI 2-sided [-2.3 to 5.3], Standard Deviation 2.38
Statistical Analysis 8: Comparison: Placebo Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.0, Standard Deviation 0.0
Statistical Analysis 9: Comparison: Any Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.9 to 0.2], Standard Deviation 1.67
Statistical Analysis 10: Comparison: Any Placebo; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 1.2, 95% CI 2-sided [-1.5 to 3.9], Standard Deviation 2.17
Statistical Analysis 11: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.5 to -0.2], Standard Deviation 1.81
Statistical Analysis 12: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.8 to 0.6], Standard Deviation 0.75
Statistical Analysis 13: Comparison: Placebo Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.0, Standard Deviation 0.0
Statistical Analysis 14: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.4 to -0.3], Standard Deviation 1.72
Statistical Analysis 15: Comparison: Any Placebo; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.4 to 0.4], Standard Deviation 0.71
Statistical Analysis 16: Comparison: Ambrisentan Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-1.2 to 0.1], Standard Deviation 1.79
Statistical Analysis 17: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 1.0, 95% CI 2-sided [-2.2 to 4.2], Standard Deviation 2.00
Statistical Analysis 18: Comparison: Placebo Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.0, Standard Deviation 0.0
Statistical Analysis 19: Comparison: Any Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Deviation 1.85
Statistical Analysis 20: Comparison: Any Placebo; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.8, 95% CI 2-sided [-1.4 to 3.0], Standard Deviation 1.79
Statistical Analysis 21: Comparison: Ambrisentan Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to 0.1], Standard Deviation 2.12
Statistical Analysis 22: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 1.0, 95% CI 2-sided [-4.5 to 6.5], Standard Deviation 3.46
Statistical Analysis 23: Comparison: Placebo Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.0, Standard Deviation 0.0
Statistical Analysis 24: Comparison: Any Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.3 to 0.3], Standard Deviation 2.30
Statistical Analysis 25: Comparison: Any Placebo; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.8, 95% CI 2-sided [-3.0 to 4.6], Standard Deviation 3.03

7. Secondary Outcome: Change From Baseline in the Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) Quality of Life (QOL) Survey Overall Score Measured at Weeks 12, 24, 36 and 48 (LOCF)
Description: The primary analysis of this secondary outcome measure is mean change from Baseline to Week 24. The changes from Baseline to Weeks 12, 36, and 48 were also evaluated. Lower scores and decreases from baseline represent improved functioning and QOL. The CAMPHOR survey was not assessed at Week 4. The total CAMPHOR score scale ranges from 0 (good) to 25 (poor). A reduction in score over time represents improvement in this patient population.
Time Frame: Baseline to Week 48
Population: All enrolled Population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 33 | 4 | 1 | 37 | 5
units on a scale
  Baseline | 8.2 (6.14) | 4.3 (5.44) | 4.0 (0.0) | 7.7 (6.12) | 4.2 (4.71)
  Week 12 | 6.8 (5.59) | 5.5 (3.11) | 2.0 (0.0) | 6.7 (5.32) | 4.8 (3.11)
  Week 24 | 7.2 (5.82) | 3.0 (2.94) | 2.0 (0.0) | 6.7 (5.69) | 2.8 (2.59)
  Week 36 | 7.7 (6.10) | 3.5 (3.70) | 3.0 (0.0) | 7.2 (5.98) | 3.4 (3.21)
  Week48 | 7.6 (6.87) | 3.8 (3.50) | 3.0 (0.0) | 7.1 (6.63) | 3.6 (3.05)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.1, 95% CI 2-sided [-2.7 to 0.4], Standard Deviation 3.98
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 1.3, 95% CI 2-sided [-6.5 to 9.0], Standard Deviation 4.86
Statistical Analysis 3: Comparison: Placebo Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -2.0, Standard Deviation 0.0
Statistical Analysis 4: Comparison: Any Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.3 to 0.6], Standard Deviation 4.09
Statistical Analysis 5: Comparison: Any Placebo; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = 0.6, 95% CI 2-sided [-4.9 to 6.1], Standard Deviation 4.45
Statistical Analysis 6: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-2.7 to 1.1], Standard Deviation 5.00
Statistical Analysis 7: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.3, 95% CI 2-sided [-7.7 to 5.2], Standard Deviation 4.03
Statistical Analysis 8: Comparison: Placebo Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -2.0, Standard Deviation 0.0
Statistical Analysis 9: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.6 to 0.9], Standard Deviation 4.84
Statistical Analysis 10: Comparison: Any Placebo; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.4, 95% CI 2-sided [-5.8 to 3.0], Standard Deviation 3.51
Statistical Analysis 11: Comparison: Ambrisentan Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.3 to 1.7], Standard Deviation 5.20
Statistical Analysis 12: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-8.1 to 6.6], Standard Deviation 4.65
Statistical Analysis 13: Comparison: Placebo Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.0, Standard Deviation 0.0
Statistical Analysis 14: Comparison: Any Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-2.2 to 1.5], Standard Deviation 5.07
Statistical Analysis 15: Comparison: Any Placebo; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-5.8 to 4.2], Standard Deviation 4.02
Statistical Analysis 16: Comparison: Ambrisentan Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.8 to 2.1], Standard Deviation 6.33
Statistical Analysis 17: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-11.4 to 10.4], Standard Deviation 6.86
Statistical Analysis 18: Comparison: Placebo Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -1.0, Standard Deviation 0.0
Statistical Analysis 19: Comparison: Any Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-2.7 to 1.9], Standard Deviation 6.28
Statistical Analysis 20: Comparison: Any Placebo; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-8.0 to 6.8], Standard Deviation 5.94

8. Secondary Outcome: Change From Baseline in World Health Organization (WHO) Functional Class (LOCF) Measured at Weeks 4, 12, 24, 36 and 48.
Description: The primary analysis of this secondary outcome measure is change from Baseline to Week 24. The changes from Baseline to Weeks 4, 12, 36, and 48 were also evaluated. WHO categories are 1 to 4 with the worst category being 4. Improvement is represented by a change in category to a lower number (for example, change from category 3 to 2), and deterioration is represented by a change in category to a higher number (for example, change from category 2 to 4). No change is represented by no change in category (for example, category 2 which remains 2).
Time Frame: Baseline to Week 48
Population: All enrolled Population
Measure: Number; unit: participants
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 33 | 4 | 1 | 37 | 5
participants
  Week 4 - Improvement | 3 | 0 | 1 | 3 | 1
  Week 4 - No Change | 29 | 4 | 0 | 33 | 4
  Week 4 - Deterioration | 0 | 0 | 0 | 0 | 0
  Week 4 - Missing Data | 1 | 0 | 0 | 1 | 0
  Week 12 - Improvement | 8 | 1 | 1 | 9 | 2
  Week 12 - No Change | 24 | 3 | 0 | 27 | 3
  Week 12 - Deterioration | 0 | 0 | 0 | 0 | 0
  Week 12 - Missing Data | 1 | 0 | 0 | 1 | 0
  Week 24 - Improvement | 12 | 2 | 1 | 14 | 3
  Week 24 - No Change | 19 | 2 | 0 | 21 | 2
  Week 24 - Deterioration | 1 | 0 | 0 | 1 | 0
  Week 24 - Missing Data | 1 | 0 | 0 | 1 | 0
  Week 36 - Improvement | 17 | 2 | 1 | 19 | 3
  Week 36 - No Change | 14 | 2 | 0 | 16 | 2
  Week 36 - Deterioration | 1 | 0 | 0 | 1 | 0
  Week 36 - Missing Data | 1 | 0 | 0 | 1 | 0
  Week 48 - Improvement | 14 | 1 | 1 | 15 | 2
  Week 48 - No Change | 17 | 3 | 0 | 20 | 3
  Week 48 - Deterioration | 1 | 0 | 0 | 1 | 0
  Week 48 - Missing Data | 1 | 0 | 0 | 1 | 0

9. Secondary Outcome: Change From Baseline in Log-transformed N-terminal Pro-B-type Natriuretic Peptide (NT-proBNP) Measured at Weeks 4, 12, 24, 36 and 48 (LOCF)
Description: The primary analysis of this secondary outcome measure is mean percent change from Baseline to Week 24. The changes from Baseline to Weeks 4, 12, 36, and 48 were also evaluated. A decrease in log-transformed measurement value (pg/mL) indicates improvement for this patient population.
Time Frame: Baseline to Week 48
Population: One patient (Any Placebo) was not evaluated for NT-proBNP. One patient (Placebo Only) had no baseline measurement, so no statistical analyses for change from baseline are given for the placebo only group (patient was only subject in this group).
Measure: Mean (Standard Deviation); unit: pg/mL (log-transformed)
Arm/Group | Ambrisentan Only | Placebo/Ambrisentan | Placebo Only | Any Ambrisentan | Any Placebo
Number analyzed (Participants) | 33 | 4 | 1 | 37 | 4
pg/mL (log-transformed)
  Baseline | 6.1 (1.10) [19.62 to 43.89] | 6.7 (1.02) [-940.3 to 93.22] | 0.0 (0.0) | 6.2 (1.10) [19.30 to 42.62] | 6.7 (1.02) [-940.3 to 93.22]
  Week 4 | 5.7 (1.02) | 6.2 (1.80) | 7.5 (0.0) | 5.7 (1.05) | 6.7 (1.46)
  Week 12 | 5.7 (1.01) | 6.3 (0.45) | 7.6 (0.0) | 5.8 (0.99) | 6.8 (0.80)
  Week 24 | 5.7 (1.03) | 6.0 (0.98) | 7.6 (0.0) | 5.7 (1.02) | 6.4 (1.12)
  Week 36 | 5.7 (1.19) | 5.9 (0.64) | 8.0 (0.0) | 5.7 (1.14) | 6.3 (1.08)
  Week 48 | 5.6 (1.16) | 6.4 (0.82) | 8.0 (0.0) | 5.7 (1.14) | 6.7 (1.01)
Statistical Analysis 1: Comparison: Ambrisentan Only; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.50
Statistical Analysis 2: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.2, Standard Deviation 0.28
Statistical Analysis 3: Comparison: Any Ambrisentan; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.49
Statistical Analysis 4: Comparison: Any Placebo; Mean change from Baseline to Week 4 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.2, Standard Deviation 0.28
Statistical Analysis 5: Comparison: Ambrisentan Only; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, Standard Deviation 0.63
Statistical Analysis 6: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.1, Standard Deviation 1.07
Statistical Analysis 7: Comparison: Any Ambrisentan; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, Standard Deviation 0.64
Statistical Analysis 8: Comparison: Any Placebo; Mean change from Baseline to Week 12 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.1, Standard Deviation 1.07
Statistical Analysis 9: Comparison: Ambrisentan Only; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.83
Statistical Analysis 10: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.7, Standard Deviation 0.34
Statistical Analysis 11: Comparison: Any Ambrisentan; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.81
Statistical Analysis 12: Comparison: Any Placebo; Mean change from Baseline to Week 24 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.7, Standard Deviation 0.34
Statistical Analysis 13: Comparison: Ambrisentan Only; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.92
Statistical Analysis 14: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, Standard Deviation 0.90
Statistical Analysis 15: Comparison: Any Ambrisentan; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.91
Statistical Analysis 16: Comparison: Any Placebo; Mean change from Baseline to Week 36 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.8, Standard Deviation 0.90
Statistical Analysis 17: Comparison: Ambrisentan Only; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.91
Statistical Analysis 18: Comparison: Placebo/Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, Standard Deviation 0.77
Statistical Analysis 19: Comparison: Any Ambrisentan; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.4, Standard Deviation 0.88
Statistical Analysis 20: Comparison: Any Placebo; Mean change from Baseline to Week 48 (LOCF); Test type: Superiority or Other; Mean Difference (Net) = -0.3, Standard Deviation 0.77

10. Secondary Outcome: Time to Clinical Worsening of PAH, Evaluated at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and After Week 48
Description: The time to clinical worsening was defined as the time from enrollment to the first occurrence of death, lung transplantation, hospitalization for PAH, atrial septostomy, or initiation of chronic parenteral prostanoid therapy. Results are presented as the Kaplan-Meier estimate (% probability) of having clinical worsening after a given time.
Time Frame: Baseline to Week 48+
Population: The Ambrisentan Only and Any Ambrisentan Groups were analyzed for Time to Clinical Worsening
Measure: Number (95% Confidence Interval); unit: Probability of clinical worsening (%)
Arm/Group | Ambrisentan Only | Any Ambrisentan
Number analyzed (Participants) | 33 | 37
Probability of clinical worsening (%)
  At Week 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 8 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 12 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 16 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 20 | 3 [0.0 to 9.1] | 3 [0.0 to 8.2]
  At Week 24 | 3 [0.0 to 9.1] | 3 [0.0 to 8.2]
  At Week 28 | 6 [0.0 to 14.7] | 6 [0.0 to 13.1]
  At Week 32 | 16 [3.1 to 29.1] | 14 [2.7 to 25.9]
  At Week 36 | 16 [3.1 to 29.1] | 14 [2.7 to 25.9]
  At Week 40 | 20 [5.6 to 34.0] | 17 [4.7 to 30.1]
  At Week 44 | 20 [5.6 to 34.0] | 17 [4.7 to 30.1]
  At Week 48 | 20 [5.6 to 34.0] | 17 [4.7 to 30.1]
  After Week 48 | 20 [5.6 to 34.0] | 17 [4.7 to 30.1]

11. Secondary Outcome: Overall Survival, Evaluated at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and After Week 48
Description: Overall survival was defined as the time from initiation of active treatment to death. Results are presented as the Kaplan-Meier estimate (% probability) of death after a given time.
Time Frame: Baseline to Week 48+
Population: The Ambrisentan Only and Any Ambrisentan Groups were analyzed for Overall Survival
Measure: Number (95% Confidence Interval); unit: Probability of death occurring (%)
Arm/Group | Ambrisentan Only | Any Ambrisentan
Number analyzed (Participants) | 33 | 37
Probability of death occurring (%)
  At Week 4 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 8 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 12 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 16 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 20 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 24 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 28 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 32 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 36 | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  At Week 40 | 4 [0.0 to 10.8] | 3 [0.0 to 9.4]
  At Week 44 | 4 [0.0 to 10.8] | 3 [0.0 to 9.4]
  At Week 48 | 4 [0.0 to 10.8] | 3 [0.0 to 9.4]
  After Week 48 | 4 [0.0 to 10.8] | 3 [0.0 to 9.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were reported through Week 48.
Description: AEs/SAEs were analyzed for patients who: received ambrisentan but not placebo ("Ambrisentan Only"); received ambrisentan and did or did not receive placebo ("Any Ambrisentan"); received placebo and did or did not receive ambrisentan ("Any Placebo"). Safety analysis was not done for the "Ambrisentan/Placebo" or "Placebo Only" groups.
Groups:
- Any Ambrisentan: Patients were assigned either ambrisentan or placebo at enrollment or randomization and received at least one dose of ambrisentan plus an approved PDE-5i
- Any Placebo: Patients were assigned placebo at randomization and received at least one dose of placebo plus an approved PDE-5i
Arm/Group | Ambrisentan Only | Any Ambrisentan | Any Placebo
Serious Adverse Events (participants affected / at risk) | 10/33 | 11/37 | 1/5
Other Adverse Events (participants affected / at risk) | 32/33 | 36/37 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan Only (N=33) | Any Ambrisentan (N=37) | Any Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 1 | 0
Right ventricular failure (Cardiac disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Gastrointestinal haemorrage (Gastrointestinal disorders) | 1 | 1 | 0
Oesophageal splasm (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 0
Chest pain (General disorders) | 1 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan Only (N=33) | Any Ambrisentan (N=37) | Any Placebo (N=5)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 3 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 2 | 0
Oedema peripheral (General disorders) | 7 | 7 | 0
Fatigue (General disorders) | 5 | 5 | 1
Chest pain (General disorders) | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 8 | 0
Urinary tract infection (Infections and infestations) | 5 | 5 | 0
Nasopharyngitis (Infections and infestations) | 3 | 4 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 3 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 0
Viral infection (Infections and infestations) | 2 | 2 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0
Brain natriuretic peptide increased (Investigations) | 3 | 3 | 0
Blood uric acid increased (Investigations) | 2 | 2 | 0
Protein total increased (Investigations) | 2 | 2 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 5 | 7 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 1
Fluid retention (Metabolism and nutrition disorders) | 3 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Headache (Nervous system disorders) | 7 | 7 | 1
Dizziness (Nervous system disorders) | 5 | 5 | 1
Carpal tunnel syndrome (Nervous system disorders) | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 10 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years